CLINICAL TRIAL: NCT02080884
Title: A MULTICENTER NON-INTERVENTIONAL STUDY EVALUATING THE BENEFIT OF THE COMBINATION OF MABTHERA (RITUXIMAB) WITH STANDARD CHEMOTHERAPEUTIC REGIMENS IN PATIENTS WITH PREVIOUSLY UNTREATED CHRONIC LYMPHOCYTIC LEUKEMIA IN HUNGARY
Brief Title: An Observational Study Examining the Effect of Added MabThera Therapy in Patients With Untreated Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29201
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CLL patients on Mabthera (rituximab)

SUMMARY:
This study will examine the effectiveness of MabThera therapy added to a standard chemotherapy regimen for the treatment of previously untreated chronic lymphocytic leukemia (CLL). Patients who have received a single prior MabThera plus chemotherapy treatment are eligible. The overall response rate of patients treated for approximately 5 months (as per current label guidelines) will be analysed according to various factors (i.e., age, concurrent treatment, and chromosomal abnormalities).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with first-line CLL having received only 1 cycle of MabThera chemotherapy
* aged >/= 18 years

Exclusion Criteria:

* Pregnant or breast-feeding
* Receipt of an investigational drug within 30 days prior to entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with untreated chronic lymphocytic leukemia (CLL)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) as assessed by the investigator using routine assessment techniques | 7 months

SECONDARY OUTCOMES:
ORR analysed according to concomitant chemotherapy | 7 months
ORR analysed according to age | 7 months
ORR analysed according to CIRS score | 7 months
ORR analysed according to certain chromosomal abnormalities | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Hungary (15):
  - Semmelweis University, First Dept of Medicine, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - Semmelweis Egyetem Aok; Iii.Sz. Belgyogyaszati Klinika, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum; III. Belgyogyaszati Klinika, Debrecen
  - Markhot Ferenc Oktato Korhaz es Rendelointezet; III. belgyogyaszat, Eger
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza; I. Belgyogyaszat-Hematologia Reszle, Gyula
  - Miskolci Semmelweis Kórház és Egyetemi Oktatókórház; Haematology Dept., Miskolc
  - Josa Andras Korhaz; Ii. Sz. Belgyogyaszati Es Haematologiai Osztaly, Nyíregyháza
  - University of Pecs, I st Dept of Internal Medicine, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ; Neurológiai Klinika, Szeged
  - Fejér Megyei Szent György Kórház; Hematologiai Osztaly, Székesfehérvár
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház; Onkológiai Osztály, Szolnok
  - Vas Megyei Markusovszky Korhaz; Haematologiai Osztaly, Szombathely
  - Szent Borbala Korhaz, Tatabanuya
  - Veszprem Megyei Csolnoky Ferenc Korhaz Nonprofit Zrt., Veszprém